CLINICAL TRIAL: NCT00802503
Title: Impact of Supplemental Parenteral Nutrition (SPN) on Infection Rate, Duration of Mechanical Ventilation and Rehabilitation in Intensive Care Unit Patients: A Quality Control Program for the Implementing of New Nutrition Guidelines
Brief Title: Impact of SPN on Infection Rate, Duration of Mechanical Ventilation & Rehabilitation in ICU Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, HEIDEGGER CP, Deputy head physician, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Protocole 07-098
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Critically Ill
Keywords: Critically ill; nutrition; randomised controlled clinical trial; human; adult; Supplemental parenteral nutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPN group (Experimental): experimental arm: Supplemental Parenteral Nutrition (SPN) is added to enteral nutrition (EN) to reach 100% of their predicted energy needs from ICU day 4.
  In the treated group, SPN is started if at day 4 energy input by EN is < 60% of energy target in order to reach 100% of energy target by peripheral or central line. Nutritional products as currently used in our institution. SPN is composed of EN and PN, both techniques being currently used in our institution.
  Interventions: Dietary Supplement: SPN
- Control gr (No Intervention): EN : start EN at 20-30 ml/h per day up to maximal 150 ml/h per day; or day1: 500 ml, day2: 1000 ml, day3: 1500 ml of EN dependant on gastrointestinal tolerance (gastric residue volume more than 500ml). Nutritional products as currently used in our institution.

INTERVENTIONS:
Dietary Supplement: SPN — SPN : in the treated group, SPN is started if at day 4 energy input by EN is < 60% of energy target in order to reach 100% of energy target by peripheral or central line.
  Arms: SPN group

SUMMARY:
Rationale: Enteral nutrition (EN) in the intensive care (ICU) patients is recommended as a standard of care. However, EN alone is often associated with insufficient energy intakes and increased complication rates. Recently the investigators proposed to decrease this deficit by combining EN and supplemental parenteral nutrition (SPN) whenever EN is insufficient (< 60% of their predicted energy needs) at day 3 after admission in the ICU.

Objective: This study aims at: a/ investigating if the delivery of optimal nutrition support (100 % of predicted energy targets) in ICU patients by the combined administration of SPN and EN optimizes their clinical outcome; b/ implementing the new ICU nutrition guidelines.

Study design: Prospective, controlled, randomized clinical study.

Study site: Service of Intensive Care, Geneva University Hospital.

Patient population: 220 ICU patients to be included: expected length of stay > 5 days, expected survival > 7 days, no contraindication to EN, obtained informed consent from themselves or their next of keen.

Exclusion criteria: refusal of consent, age < 18 years, short bowel syndrome, significant persistent gastrointestinal dysfunction with ileus, high output proximal fistula (> 1,5 liter/d), patients receiving PN.

Nutrition: At day 3 after admission, if energy input is < 60%; patients are randomized into either the "Control group" (EN alone) or the "SPN group" (EN + PN) to reach 100% of their predicted energy needs. Tight glycaemic control (target 6.0 to 8.3 mmol/l) to be achieved according to our local practice by insulin administration.

Study endpoints:

* Primary: nosocomial infections (CDC criteria)
* Secondary: Mechanical ventilation duration, ICU and hospital length of stay, antibiotic free days, ICU complications (extra-renal epuration, neurological, cardiac and respiratory complications), energy and protein balance, 28 days clinical outcome.

DETAILED DESCRIPTION:
Introduction:

Nutritional support of the intensive care (ICU) patients is recommended as a standard of care. It is also strongly recommended to start enteral feeding as soon as possible whenever the gastrointestinal tract is functioning (1). However, studies have repeatedly shown that with enteral support alone, insufficient energy and protein intakes often occur (2). The resulting energy and protein deficit is associated with an increased complication rate in ICU patients (3-5). Recently we proposed to decrease this deficit by promoting a combined nutrition support by enteral nutrition (EN) and supplemental parenteral nutrition (SPN) whenever EN is insufficient (6).

Contrary to former beliefs, recent meta-analyses show that parenteral nutrition (PN) does not carry excess mortality (7, 8). These reports convey a concept that is a major break-through in current routine of nutritional support in ICU patients by promoting a much wider use of PN. SPN could be the optimal modality to provide the calculated energy targets if this cannot be reached by EN alone. To improve ICU patient's outcome and minimise complications, we propose to implement feeding protocols which combine both EN and PN, when EN is insufficient to cover more than 60% of caloric needs at day 4 to reach 100% of the energy targets by adding PN from day 4 (6).

Hypothesis:

The administration of SPN, in ICU patients receiving < 60% of targeted energy needs by EN alone, has a positive impact on their clinical outcome by optimising their nutritional support (reduced infectious complications rate, mechanical ventilation days, duration of ICU and hospital length of stay and rehabilitation).

Objective:

The aim of the present study is to investigate if the delivery of optimal nutrition support (100 % of predicted energy targets) in ICU patients achieved with the combined administration of SPN and EN optimizes their clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Expected ICU stay > 5 days
* Expected survival > 7 days
* No contraindication to EN
* Obtained informed consent

Exclusion Criteria:

* Refusal of consent
* Age < 18 years
* Short bowel syndrome
* Significant persistent gastrointestinal dysfunction with ileus
* High output proximal fistula (> 1.5 liter/d)
* Patients receiving PN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia P HEIDEGGER, MD, Principal Investigator — Division of Intensive Care, 1211 Geneva 14, Switzerland
Locations (2):
- Switzerland (2):
  - Service of Intensive Care, Geneva University Hospital,, Geneva
  - Service de Médecine Intensive Adulte et Centre des Brûlés, Lausanne

REFERENCES:
- [Background] Heidegger CP, Romand JA, Treggiari MM, Pichard C. Is it now time to promote mixed enteral and parenteral nutrition for the critically ill patient? Intensive Care Med. 2007 Jun;33(6):963-9. doi: 10.1007/s00134-007-0654-7. Epub 2007 Apr 28. PMID 17468845
- [Derived] Heidegger CP, Berger MM, Graf S, Zingg W, Darmon P, Costanza MC, Thibault R, Pichard C. Optimisation of energy provision with supplemental parenteral nutrition in critically ill patients: a randomised controlled clinical trial. Lancet. 2013 Feb 2;381(9864):385-93. doi: 10.1016/S0140-6736(12)61351-8. Epub 2012 Dec 3. PMID 23218813

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: EN : start EN at 20-30 ml/h per day up to maximal 150 ml/h per day; or day1: 500 ml, day2: 1000 ml, day3: 1500 ml of EN dependant on gastrointestinal tolerance (gastric residue volume more than 500ml). Nutritional products as currently used in our institution.
- SPN Group: experimental arm: Supplemental Parenteral Nutrition (SPN) is added to enteral nutrition (EN) to reach 100% of their predicted energy needs from ICU day 4.
  In the treated group, SPN is started if at day 4 energy input by EN is < 60% of energy target in order to reach 100% of energy target by peripheral or central line. Nutritional products as currently used in our institution. SPN is composed of EN and PN, both techniques being currently used in our institution.
  SPN : SPN : in the treated group, SPN is started if at day 4 energy input by EN is < 60% of energy target in order to reach 100% of energy target by peripheral or central line.
Period: Overall Study
Arm/Group | Control Group | SPN Group
Started | 152 | 153
Completed | 142 | 133
Not Completed | 10 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control gr | SPN Group | Total
Number analyzed (Participants) | 152 | 153 | 305
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 83 | 174
  >=65 years | 61 | 70 | 131
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (16) | 61 (16) | 60 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 90
  Male | 105 | 110 | 215
Region of Enrollment [Number; unit: participants]
  Switzerland | 152 | 153 | 305

OUTCOME MEASURES:

1. Primary Outcome: Documented Infection Rate
Description: Infection, defined according to CDC criteria during the ICU and hospital stay, occurrence between day 9 and day 28
Time Frame: 20 days
Measure: Number; unit: Infections
Groups:
- Control gr: EN : start EN at 20-30 ml/h per day up to maximal 150 ml/h per day; or day 1: 500 ml, day 2: 1000 ml, day 3: 1500 ml of EN dependent on gastrointestinal tolerance (gastric residue volume more than 500 ml). Nutritional products as currently used in our institution.
Arm/Group | Control gr | SPN Group
Number analyzed (Participants) | 152 | 153
Infections | 58 | 41

2. Secondary Outcome: Hours on Mechanical Ventilation in All Patients
Description: Mechanical ventilation hours during study duration (days 1-28)
Time Frame: 28 days
Population: The intention to treat analysis included all patients randomly assigned to the intervention SPN group (153) or control group EN (152). The per protocol analysis included only patients who fully completed the 5-day intervention in the ICU (SPN group(133); EN group (142).
Measure: Mean (95% Confidence Interval); unit: hours of mechanical ventilation
Arm/Group | Control gr | SPN Group
Number analyzed (Participants) | 152 | 153
hours of mechanical ventilation | 166 [138 to 189] | 153 [126 to 178]

3. Secondary Outcome: Antibiotic Free Days
Description: Number of days between day 9 to day 28 (follow-up period) free of antibiotics
Time Frame: 20 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: number of days
Arm/Group | Control gr | SPN Group
Number analyzed (Participants) | 152 | 153
number of days | 12 [10 to 13] | 14 [12 to 15]

4. Secondary Outcome: Total Energy Intake During the Intervention Period , Between Day 4 and Day 8.
Description: Percentage of energy target; in the SPN group the goal was to achieve 100% of the energy target during intervention (day 4 to day 8.The energy target was measured by indirect calorimetry in 198 patients of 305(65%),otherwise energy target was calculated by 25 kcal per kg of ideal body weight for women and 30 kcal per kg of ideal body weight for men and anamnestic body weight was used for patients with a body mass index of 20 kg/m2 or lower.
Time Frame: 5 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of energy target
Arm/Group | Control gr | SPN Group
Number analyzed (Participants) | 152 | 153
% of energy target | 77 (27) | 103 (18)

5. Secondary Outcome: General Mortality
Time Frame: 28 days
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Control Group: EN : start EN at 20-30 ml/h per day up to maximal 150 ml/h per day; or day 1: 500 ml, day 2: 1000 ml, day 3: 1500 ml of EN dependent on gastrointestinal tolerance (gastric residue volume more than 500 ml). Nutritional products as currently used in our institution.
Arm/Group | Control Group | SPN Group
Number analyzed (Participants) | 152 | 153
participants | 28 (18) [13 to 25] | 20 (13) [9 to 19]

6. Secondary Outcome: Days in ICU
Description: Days in ICU
Time Frame: 28 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: days in ICU
Arm/Group | Control gr | SPN Group
Number analyzed (Participants) | 152 | 153
days in ICU | 13 [12 to 14] | 13 [11 to 14]

7. Secondary Outcome: ICU Mortality
Time Frame: 28 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Control gr | SPN Group
Number analyzed (Participants) | 152 | 153
participants | 12 [5 to 13] | 8 [3 to 10]

8. Secondary Outcome: Protein Delivery During the Intervention Period From Day 4 to Day 8
Description: Percentage of protein target between day 4 to 8. Protein target was set to 1.2 g per kg of ideal body weight a day.
Time Frame: 5 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of protein target
Groups:
- Controle gr: EN : start EN at 20-30 ml/h per day up to maximal 150 ml/h per day; or day 1: 500 ml, day 2: 1000 ml, day 3: 1500 ml of EN dependent on gastrointestinal tolerance (gastric residue volume more than 500 ml). Nutritional products as currently used in our institution.
- SPN gr: experimental arm: Supplemental Parenteral Nutrition (SPN) is added to enteral nutrition (EN) to reach 100% of their predicted energy needs from ICU day 4.
  In the treated group, SPN is started if at day 4 energy input by EN is < 60% of energy target in order to reach 100% of energy target by peripheral or central line. Nutritional products as currently used in our institution. SPN is composed of EN and PN, both techniques being currently used in our institution.
  SPN : SPN : in the treated group, SPN is started if at day 4 energy input by EN is < 60% of energy target in order to reach 100% of energy target by peripheral or central line.
Arm/Group | Controle gr | SPN gr
Number analyzed (Participants) | 152 | 153
percentage of protein target | 71 (27) | 100 (16)

9. Secondary Outcome: Days in Hospital
Description: hospital length of stay
Time Frame: 28 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: days in hospital
Arm/Group | Control gr | SPN Group
Number analyzed (Participants) | 152 | 153
days in hospital | 32 [29 to 39] | 31 [29 to 38]

ADVERSE EVENTS:
Time Frame: The follow up period was until day 28.
Description: No adverse events were observed during the intervention period from day 4 to day 8.
Arm/Group | Control gr | SPN Group
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/153
Other Adverse Events (participants affected / at risk) | 0/152 | 0/153

LIMITATIONS AND CAVEATS:
The trial was limited by the fact that it was not double blinded by design. However, the risk of bias was reduced because the investigators worked independently from the physicians in charge of the patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No